CLINICAL TRIAL: NCT01632735
Title: Mobile Continuing Care Approach for Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azusa Pacific University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5K01DA027754-03 (NIH); 1K01DA027754-01A1 (NIH)
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-07

CONDITIONS: Addiction
Keywords: Continuing Care; Youth Substance Abuse; Recovery Support; Mobile Texting
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile Continuing Care (Experimental): Behavioral: 12-week Structured Texting intervention focused on recovery monitoring, feedback for self-management, social support and education
  Interventions: Behavioral: Mobile Continuing Care
- Standard Continuing Care as Usual (No Intervention): Continuing care as usual to 12-step facilitation (Anonymous group)

INTERVENTIONS:
Behavioral: Mobile Continuing Care — Behavioral: Mobile Texting 12-week intervention. Delivers daily Recovering monitoring, self-management feedback, and education/social support
  Arms: Mobile Continuing Care

SUMMARY:
The primary purpose of this study is to test the effectiveness of a pilot mobile based continuing care program (monitoring/feedback texting) relative to standard continuing care as usual in reducing relapse and improving psychosocial functioning outcomes in a youth population (under 24) with substance abuse problems.

DETAILED DESCRIPTION:
This study will include approximately 80 participants randomized to either 12 weeks of mobile continuing care (intervention) or standard continuing care as usual (control). Participants will be recruited from the treatment programs in Los Angeles County, including Matrix Institute on Addictions, Tarzana Treatment, Twin Town, Phoenix House, and Cri-Help. During the 12-week active program, participants will be monitored monthly via telephone data collection. Both groups will be followed for 10-months using repeated assessments (self-report and urine specimens) at baseline (month 0) and at follow-up points (months 3, 6, and 9).

ELIGIBILITY:
Inclusion Criteria:

1. Youth between 12 and 24 years old
2. Youth in treatment for substance abuse
3. Youth who complete treatment (minimum 12 weeks)
4. Youth who have the cognitive capacity to understand study procedures and agree to participate

Exclusion Criteria:

1. Presence of an adverse (life threatening) medical condition that could interfere with study participation.
2. Presence of psychiatric co-occurring illness or symptoms warranting safety concerns or continued treatment, including acute suicide risk; and
3. Current homelessness (unless residing in recovery home for which contact information can be provided).

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Gonzales-Castaneda, MPH, PhD, Principal Investigator — Azusa Pacific University
Locations (1):
- Azusa Pacific University Psychology Department, Azusa, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Continuing Care as Usual: Continuing care as usual (12-step facilitation) group
Period: Overall Study
Arm/Group | Mobile Continuing Care | Standard Continuing Care as Usual
Started | 40 | 40
Completed | 36 | 37
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Population: This study included 80 substance abusing youth who completed treatment and participated in a pilot aftercare project called Project ESQYIR (Educating & Supporting inquisitive Youth in Recovery). Youth were randomized to the mobile aftercare intervention (n=40) or aftercare as usual control (n=40).
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Continuing Care | Standard Continuing Care as Usual | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (3.1) | 19.0 (3.1) | 20.4 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 25 | 32 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 20 | 30
  Not Hispanic or Latino | 30 | 20 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 22 | 12 | 34
  More than one race | 10 | 20 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
education [Mean (Standard Deviation); unit: years] | 14.0 (2.3) | 12.0 (2.0) | 12.9 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Primary Substance Use (Defined as Substance Received Treatment for)
Description: Primary substance use relapse was measured by urine tests (0 = negative, 1 = positive).
Time Frame: Baseline, discahrge, 3 month follow-up, 6 month follow-up, 9 month follow-up
Population: An intent to treat model was used. The primary outcome measure is primary substance use measured by urine drug test at baseline, discharge as well as at 3-, 6-, and 9-month follow-ups. Study retention at discharge was 95%, 92.5% at 3 months, 86.2% at 6 months, and 82.5% at 9 months.
Measure: Number; unit: percentage of positive urines
Arm/Group | Mobile Continuing Care | Standard Continuing Care as Usual
Number analyzed (Participants) | 40 | 40
percentage of positive urines
  baseline substance use | 47.5 | 41.5
  discharge substace use | 14.7 | 62.9
  3-month follow-up substace use | 21.4 | 59.3
  6-month follow-up substace use | 16.7 | 50.0
  9-month follow-up substace use | 11.1 | 14.3
Statistical Analysis 1: Comparison: Mobile Continuing Care vs Standard Continuing Care as Usual; Test type: Superiority or Other; p < 0.05, GEE; Generalized Estimating Equations regression examined primary relapse (measured by urinalysis) over time by condition, controlling for age and gender; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.57 to 0.99]

2. Secondary Outcome: Participation in Recovery Behaviors Over Time
Description: Recovery behaviors defined as mean number of days doing extracurricular/recovery-goal directed activities using repeated measures over time.
Time Frame: baseline, discharge, 3-, 6- and 9-month follow-ups
Population: Intent to treatment model was used. Mixed modeling used to examine differences in recovery behaviors (measured by mean days doing extracurricular/recovery-goal directed activities) over time between study conditions.
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Mobile Continuing Care | Standard Continuing Care as Usual
Number analyzed (Participants) | 40 | 40
days per month
  baseline recovery behaviors | 12.1 (9.7) | 14.5 (11.7)
  discharge recovery behaviors | 17.3 (8.5) | 10.3 (11.4)
  3-month recovery behaviors | 14.5 (9.5) | 11.97 (11.96)
  6-month recovery behaviors | 17.5 (10.6) | 13.8 (12.9)
  9-month recovery behaviors | 18.4 (10.6) | 12.4 (16.6)
Statistical Analysis 1: Comparison: Mobile Continuing Care vs Standard Continuing Care as Usual; Mixed modeling using a repeated-measures random-effects model was conducted to test for the effects of treatment (dummy coded with 1 = mobile intervention, 0 = control) and time as well as the treatment x time interaction on the primary outcome measures of recovery behaviors mean days over time (baseline, discharge, 3, 6, and 9-month follow-ups); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Analyses controlled for age and gender; Beta (timexcondition) = 0.239, 95% CI 2-sided [0.219 to 0.248]

3. Secondary Outcome: Recovery Confidence (Self-efficacy) Over Time
Description: Change/improvements in mean recovery confidence score over time (measured by question "How confident are you in your ability to be completely abstinent (clean) from alcohol and drugs in the next 30 days?" (units on scale included 0=not at all, 1=slightly, 2=moderately, 3=considerably, 4-extremely).
Time Frame: baseline, discharge, 3-, 6-, and 9-month follow-ups
Population: Used an intent to treat design. Examined the effects of the intervention (mobile continuing care) compared to aftercare as usual on change in recovery self-confidence over time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Continuing Care | Standard Continuing Care as Usual
Number analyzed (Participants) | 40 | 40
units on a scale
  baseline confidence rating | 2.40 (1.3) | 2.53 (1.2)
  discharge confidence rating | 2.73 (1.03) | 2.57 (1.5)
  3-month follow-up confidence rating | 2.67 (1.3) | 2.43 (1.4)
  6-month follow-up confidence rating | 3.20 (1.02) | 2.51 (1.50)
  9-month follow-up confidence rating | 2.85 (1.3) | 2.73 (1.3)
Statistical Analysis 1: Comparison: Mobile Continuing Care vs Standard Continuing Care as Usual; Mixed modeling using a repeated-measures random-effects model was conducted to test for the effects of treatment (dummy coded with 1 = mobile intervention, 0 = control) and time as well as the treatment x time interaction on the outcome measure of recovery confidence mean score over time; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; A repeated-measures model tested for effects of treatment vs. control on recovery self-confidence over time controlling for age and gender; Beta (time x condition) = 0.115, 95% CI 2-sided [0.106 to 0.123]

4. Secondary Outcome: Social Support Utilization
Description: Self-help utilization was measured by the question: "In the past 30 days, how many days did you attend self-help meetings like AA or NA to support your recovery?"
Time Frame: Baseline, discahrge, 3 month follow-up, 6 month follow-up, 9 month follow-up
Population: Intent to treat model was used to assess the effects of the intervention (mobile continuing care) compared to aftercare as usual in terms of improvements in social support service utilization over time (baseline, discharge and follow-ups: 3-, 6- and 9-months post-discharge).
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Mobile Continuing Care | Standard Continuing Care as Usual
Number analyzed (Participants) | 40 | 40
days per month
  baseline social support utilization | 12.8 (10.3) | 9.8 (8.1)
  discharge social support utilization | 8.6 (10.1) | 2.8 (6.6)
  3-month follow-up social support utilization | 7.4 (9.5) | 2.4 (6.0)
  6-month upport utilization | 6.1 (8.5) | 2.8 (7.3)
  9-month upport utilization | 4.9 (7.7) | 2.8 (7.2)
Statistical Analysis 1: Comparison: Mobile Continuing Care vs Standard Continuing Care as Usual; Mixed modeling using a repeated-measures random-effects model was conducted to test for the effects of treatment (dummy coded with 1 = mobile intervention, 0 = control) and time as well as the treatment x time interaction on the outcome measure of self-help utilization (mean days in past month) over the study period (baseline, discharge, and 3-, 6-, and 9-month follow-ups); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Analyses controlled for age and gender; Beta effect (timexcondition) = 0.217, 95% CI 2-sided [0.2 to 0.233]

ADVERSE EVENTS:
Time Frame: During the 9-month study period.
Description: Serious and non-serious adverse events were not observed during the study period.
Arm/Group | Mobile Continuing Care | Standard Continuing Care as Usual
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
Pilot study limiting number of participants recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No